CLINICAL TRIAL: NCT05951335
Title: Effectiveness of m-Health Supportive Care Transition Program in Improving Post-Discharged Outcomes Among Traumatic Brain Injury Caregivers: A Randomized Controlled Trial
Brief Title: m-Health Supportive Care Transition Program in Improving Post-Discharged Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Amelia Ganefianty, Principal Investigator, Prince of Songkla University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: AG2023
Record Dates: First submitted 2023-07-03; First posted 2023-07-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Traumatic Brain Injury; Caregiver Burden; Stress
Keywords: m-health; Burden; Stress transition; Transitional care
MeSH Terms: conditions — Brain Injuries, Traumatic; Caregiver Burden

STUDY DESIGN:
Intervention Model Description: In cross-study, study participants will be transferred to all treatment groups (both test and reference formulations) after the study period is over. Being a collection of the same population, the advantage of the cross-study was that the patients acted as their controls.
Who Masked: Outcomes Assessor
Masking Description: In this study, the coding process and statistical analysis will carry out by third parties (statisticians) to reduce bias in the results and conflicts of interest.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The group who received The m-Health supportive care transition program consists of education and providing face-to-face information assisted by an android-based application that can access via a smartphone, skill demonstration, assessment of the readiness of hospital discharge, as well as weekly monitoring and follow-up after the patient is discharged from the hospital. This application provides education and information on TBI caregivers regarding (a) how to treat patients with TBI at home, which includes wound care and how to provide nutrition, (b) recognize signs of infection in wounds of craniotomy, (c) recognize emergencies in cases of TBI patients at home, (d) stress management, and (e) how to arrange a schedule for the care of patients with TBI at home. This program complements routine care, including education about physical health, TBI medical problems, and how to treat TBI patients at home.
  Interventions: Other: m-Health Transition Care Program
- Control group (No Intervention): The group who received the usual care from nurses for the caregiver-patient with TBI in the ward before discharge from the hospital consists of education about physical health and TBI medical problems and how to treat TBI patients at home. This includes wound care education, medication administration, and schedule control at the hospital after patients with TBI go home. After discharge, there is no program carried out by nurses.

INTERVENTIONS:
Other: m-Health Transition Care Program — The m-Health supportive care transition program is a routine support program for caregivers of TBI patients. This program consists of education and providing face-to-face information assisted by an android-based application that can access via a smartphone, skill demonstration, assessment of the readiness of hospital discharge, as well as weekly monitoring and follow-up after the patient is discharged from the hospital. This application provides education and information on TBI caregivers regarding (a) how to treat patients with TBI at home, which includes wound care and how to provide nutrition, (b) recognize signs of infection in wounds of craniotomy, (c) recognize emergencies in cases of TBI patients at home, (d) stress management, and (e) how to arrange a schedule for the care of patients with TBI at home. This program complements routine care, which consists of education about physical health, TBI medical problems, and how to treat TBI patients at home.
  Arms: Intervention group

SUMMARY:
This intervention study aims to investigate the effects of the m-Health supportive care transition program on response patterns (transition stress and the burden of caregiving) among traumatic brain injury (TBI) caregivers and patients' readmission rate one month after hospital discharge. Specific objectives:

1. Compare the response patterns (transition stress and the burden of caregiving) of TBI caregivers before and after receiving the program within the group.
2. Compare TBI caregivers' response patterns (transition stress and the burden of caregiving) between the control and intervention groups.
3. Compare patients' readmission rates at one month after hospital discharge between the control and intervention groups

TBI caregivers are divided into two groups: the intervention group (who receive the transitional care program) and the control group (who receive the standard care program) according to standard operating procedures applicable in the hospital.

If there is a comparison group: Researchers will compare [insert groups] to see if [insert effects]

DETAILED DESCRIPTION:
The M-health Program Application prototype concept is designed to assist the need for intervention in providing patient care during the transition of patients with TBI from hospital care to home, which nurses and patients can use as users. This program begins with education and face-to-face information using flipcharts and direct demonstration skills. The application can provide an overview of interventions carried out by TBI caregivers while at home. This will later improve the quality of service in the rehabilitation of post-TBI. This application provides education and information on TBI caregivers regarding (a) how to treat patients with TBI at home, which includes craniotomy wound care and how to provide nutrition, (b) recognize signs of infection in wounds of craniotomy, (c) recognize emergencies in cases of TBI patients at home, (d) stress management, and (e) how to arrange a schedule for the care of patients with TBI at home. This program complements routine care, including education about physical health, TBI medical problems, and how to treat TBI patients at home.

When patients with TBI are still being treated at the hospital, researchers will directly educate TBI caregivers about the components contained in m-Health. M-Health is a caregiver-assisting tool in remembering educational materials provided by researchers while in the hospital so that TBI caregivers can access educational materials quickly accompanied by educational videos that can make it easier for them to treat patients with TBI at home. There is also an online chat service within m health that allows direct chat communication between researchers and caregivers at home and can facilitate researchers in ensuring that caregivers use m-health at home. There is also a feature that provides a contact number that can be contacted when the caregiver has problems or needs assistance in caring for patients at home.

The m-Health program is also accompanied by monitoring and follow-up telephones to support TBI caregivers and assist in solving TBI caregivers' problems during the transition from hospital to home. M-health Program Application is run using an Android-based operating system. Android is software used by mobile devices that includes an operating system, middleware, and critical applications. Application development on the Android platform uses the Framework Flutter programming language. In addition, Android relies on Linux version 2.6 for core system services such as security, memory management, process management, network stack, and driver models. The kernel also acts as an abstraction layer between the hardware and the rest of the software stack.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Family members who identify themselves as responsible persons in caring for patients at home or primary caregivers who other family members have assigned to care for patients
* Caregivers who provide care for patients with moderate or severe traumatic brain injury (TBI)
* Able to communicate, read, write, and speak Indonesian well
* Willing to be involved in research; Have an Android phone and can operate it well
* Has a measurement score of The Preparedness for Caregiving Scale (PCS) <16

Exclusion Criteria:

* Caregivers for patients with TBI with comorbidity (heart disorders, kidney disorders, and diabetes mellitus).
* Caregivers for TBI patients who will move locations outside of West Java Province after hospitalization or are sick at the hospital also not be included in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Readiness of hospital discharge used The Preparedness for Caregiving Scale (CPS) | 5 weeks
  the state and process of caregivers for patients with TBI who are characterized by physical stability and competence to manage the care of patients with TBI at home, adequate support for coping after leaving the hospital, psychological ability to care for patients at home, and having sufficient information and knowledge. to address common problems in patients with TBI. There are 8 question items. Responses are rated on a 5 point scale with scores ranging from 0 (not at all prepared) to 4 (very well prepared). The scale is scored by calculating the mean of all items answered with a score range of 0 to 4. If the total score is less than 16, it is indicated that the caregiver is not ready for hospital discharge. Still conversely, if the total score is more than 16, the caregiver is ready for hospital discharge.
Stress transition used the Caregiver Stress Self-Assessment | 5 weeks
  as a demand in which TBI caregivers do not have automatic adaptive responses when facing phases of care for patients with TBI in different settings, from hospital to home. Questionnaire containing a list of 20 statements. After each statement, indicate how often you feel that way: never, rarely, sometimes, quite frequently, or nearly always. The answer scores are Never = 0, Rarely = 1, Sometimes = 2, Quite Frequently = 3 Nearly always = 4. Total scores will be summary.
Caregiver burden used the Short- Zarit Burden Interview (ZBI) | 5 weeks
  the level of multifaceted tension felt by caregivers caring for patients with TBI at home after discharge from the hospital, related to caregiver health, psychological well-being, finances, social presence, and relationships between caregivers and patients. The Short- Zarit Burden Interview (ZBI) is a 12-item instrument for measuring the caregiver's perceived burden of providing family care. The 12 items are assessed on a 5-factor Likert scale. Items 1 to ten have positive statements so that the value ranges from 0 = 'never' to 4 = 'nearly continually.' While items number 11 and 12 have negative questions, the value ranges from 0 = 'nearly continually' to 4 = 'never. ' Item ratings are introduced to give a complete rating ranging from 0 to 48, with higher scores indicating extra burden.

SECONDARY OUTCOMES:
Readmission rate used hospital's medical record database | 5 weeks
  the subsequent inpatient admission of a patient with TBI to an acute care facility at least 30 days after discharge of the date of discharge from the hospital

CONTACTS AND LOCATIONS:
Locations (1):
- Amelia Ganefianty, Songkhla, Thailand

IPD SHARING:
Plan to Share IPD: No